CLINICAL TRIAL: NCT03777046
Title: Addressing Maternal Mental Health Needs During Pediatric Acute Care Hospitalizations
Brief Title: Maternal Mental Health in the Hospital Setting
Acronym: MMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michelle Lopez (Other)
Responsible Party: Sponsor-Investigator, Michelle Lopez, Principal Investigator, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H44040
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Post Partum Depression
Keywords: PPD; Post Partum; Post Partum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Screen fail subjects (No Intervention): Mothers and their babies that meet inclusion criteria for the study, but score less than 10 on the Edinburgh Postpartum Depression Scale (EPDS)
- PPD Control subjects (Active Comparator): Mothers and their babies that meet inclusion criteria for the study, that score 10 or more on the Edinburgh Postpartum Depression Scale (EPDS) that will receive Standard of care treatment. SOC treatment includes social work consult with information about follow up options for PPD.
  Interventions: Behavioral: Standard of Care (SOC)
- PPD Intervention subjects (Experimental): Mothers and their babies that meet inclusion criteria for the study, that score 10 or more on the Edinburgh Postpartum Depression Scale (EPDS) that will receive the experimental intervention. Intervention includes SOC treatment as well as psychology therapy (CBT) in the hospital.
  Interventions: Behavioral: SOC with Psychology Therapy (CBT)

INTERVENTIONS:
Behavioral: Standard of Care (SOC) — Mothers that meet inclusion criteria for the study, that score 10 or more on the Edinburgh Postpartum Depression Scale (EPDS) that will receive Standard of care treatment. SOC treatment includes social work consult with information about follow up options for PPD.
  Arms: PPD Control subjects
Behavioral: SOC with Psychology Therapy (CBT) — Mothers that meet inclusion criteria for the study, that score 10 or more on the Edinburgh Postpartum Depression Scale (EPDS) that will receive the experimental intervention. Intervention includes SOC treatment as well as psychology therapy (CBT) in the hospital.
  Arms: PPD Intervention subjects

SUMMARY:
Perinatal (around the time of birth) mental health disorders are common difficulties of pregnancy. Perinatal depression is made up of major and minor depressive events during pregnancy and the first 12 months after delivery. It is estimated that 11%-19% of mothers suffer from perinatal depression. However, rates may be significantly higher among some subpopulations.

Left untreated, post partum depression (PPD) is linked with several significant negative health impacts on the mother, her infant, and their families. PPD is linked with lower quality maternal-child relationship, and this change in emotional attachment can lead to physiologic changes and poorer cognitive outcomes in the infant.

The purpose of this study is to determine the maternal mental health effect of postpartum depression screening and intervention during infants' short term hospitalizations. The study is also aiming to define effects of PPD short term hospitalization interventions on maternal PPD follow up and child health based on well child care (WCC), emergency department (ED) visits, hospital readmissions, and parent's feelings on child's health.

DETAILED DESCRIPTION:
Study participants will complete a survey about their general needs and access to resources and a survey to screen for postpartum depression to determine if the participant will be enrolled. Based on the answers provided, the study team may recommend that the participant seek additional medical care, and may notify the participant's doctor, the child's doctor, and hospital officials if the study team believes that the participant needs further medical care for depression.

Half of the study participants will receive a social work consult and treatment with psychology therapy in the hospital. The psychology therapy will be 2-3 fifty-minute therapy sessions while the child is in the hospital. An outpatient psychiatry/psychology follow up appointment will be offered if needed as per routine care.

Discharge Follow Up:

A discharge follow up questionnaire and survey will be completed on an electronic tablet around the time of the baby's discharge home from the hospital or within 1 week of being at home. The survey can be completed over the phone or it can be sent via email or text to complete the survey online.

One Month Follow Up:

A one-time follow up questionnaire and survey will be completed 1 month after discharge from the hospital. The survey can be completed in approximately 5 - 10 minutes over the phone or it can be sent via email or text to complete the survey online.

The other half of the study participants will receive social work consult with information about follow up options for PPD per current standard of care for mothers identified as having postpartum depression in the hospital setting.

As part of this study a review of the child's medical record, including data collection, will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years old.
2. Mothers of infants ≤365 days of age admitted to the acute care floors at Texas Children's Hospital Medical Center Campus and their infant based on date of birth in Epic.
3. English or Spanish speaking mother.
4. Willing and able to provide informed consent.
5. Mothers with Edinburgh Postpartum Depression Scale (EPDS) score more than or equal to 10
6. Ability to complete study protocol.

NOTE: Inclusion item # 3 is as per their choice for bilingual mothers.

Exclusion Criteria:

1. Mother and infant(s) reside outside 50-mile radius of Texas Children's Hospital Medical Center Campus based on address on demographic form.
2. Mother is not the primary caregiver of infant(s) confirmed at time of informed consent.
3. Enrollment in this study during previous hospitalization based on duplicate identified in database.
4. Currently under care of psychiatrist or psychologist as reported in screening questionnaire.

NOTE: Exclusion item #2 is self-reported by the mothers at the time of screening for eligibility for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on the population being studied, only females with children that have given birth will be included.
Enrollment: 545 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Difference in PPD score | at Month 1
  PPD score will be measured using the Edinburgh Postnatal Depression Scale (EPDS). A score less than 8 suggests depression is not likely. A score of 9-11 suggests depression is possible. A score of 12-13 indicates fairly high possibility of depression. A score of 14 and higher suggest probable depression. Positive score of 1, 2 or 3 on question 10 suggests there is a suicidality risk.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Lopez, MD, Principal Investigator — Texas Children's Hospital/Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital - Women's Pavilion, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No